CLINICAL TRIAL: NCT02864524
Title: Effects of Manipulative Therapy in the Lower Thoracic and Cervical Spine in Subjects With Fibromyalgia Syndrome
Brief Title: Manipulative and Massage Therapy in the Lower Thoracic and Cervical Spine in Subjects With Fibromyalgia Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-499
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Fibromyalgia
Keywords: Physical Therapy Modalities; Exercises; Musculoskeletal Manipulations
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Massage; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manipulative and Massage Therapy (Experimental): Ten sessions (2/week):
  * High speed and low amplitude technique to lower cervical spine (C3-C4).
  * Dog technique flexion for high thoracic area (T1-T4).
  * Dog technique flexion for mid-thoracic area (T5-T8).
  * Dog technique flexed to low thoracic (T6-T12).
  Classic Massage Therapy during 40 minutes (2 time / week):
  Interventions: Other: Manipulative and Massage Therapy
- Exercise Program (Active Comparator): Ten sessions (2 time/ week): Initial heating and continuing with aerobic and muscle stretching exercises.
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Manipulative and Massage Therapy
  Arms: Manipulative and Massage Therapy
Other: Exercise Program
  Arms: Exercise Program

SUMMARY:
Objective: Compare degree of improvement can reach patients diagnosed with fibromyalgia syndrome, by treatment with Manipulative and Massage Techniques versus an exercise program for lower thoracic and cervical spine.

Study Design: A single-blind randomized controlled trial was conducted on patients with fibromyalgia syndrome (FMS).

Setting: Clinical setting. Methods: Sixty-four subjects with FMS were randomly assigned to an experimental group receiving manipulative and massage therapy, or to a control group for exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Fibromyalgia Syndrome.
* Limitation of usual activities due to pain on at least 1 day in the previous 30 days.
* Agreement to attend evening therapy sessions.
* Non-practice of regular physical activity.

Exclusion Criteria:

* A history of surgery.
* The presence of comorbid conditions (e.g., morbid obesity, inflammatory diseases, irritable bowel syndrome and interstitial cystitis).
* A history of whiplash injury.
* Severe physical disability.
* Uncontrolled endocrine disorders (e.g., hyperthyroidism, diabetes).
* Illness (e.g., schizophrenia or substance abuse).
* The use of medication other than as-needed analgesics (excluding long-term narcotics).
* Malignancy.
* Psychiatric disorders.
* A score of ≥ 9 points in the Beck depression inventory.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-11 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Changes from Baseline, and 5 weeks
  A 10-point numerical scale (0 = no pain, 10: very severe pain)

SECONDARY OUTCOMES:
McGill Pain Questionnaire | Changes from Baseline, and 5 weeks
Pittsburgh Quality of Life Questionnaire | Changes from Baseline, and 5 weeks
Quality of Life Questionnaire (SF-36) | Changes from Baseline, and 5 weeks
Fibromyalgia Impact Questionnaire (FIQ) | Changes from Baseline, and 5 weeks
Hospital Anxiety and Depression Scale (HADS) | Changes from Baseline, and 5 weeks
Beck Depression Inventory | Changes from Baseline, and 5 weeks
Fatigue Impact Scale (FIS) | Changes from Baseline, and 5 weeks
Schöber Test | Changes from Baseline, and 5 weeks
Pressure Algometry | Changes from Baseline, and 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaida María Castro-Sánchez, Almería, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ericsson A, Palstam A, Larsson A, Lofgren M, Bileviciute-Ljungar I, Bjersing J, Gerdle B, Kosek E, Mannerkorpi K. Resistance exercise improves physical fatigue in women with fibromyalgia: a randomized controlled trial. Arthritis Res Ther. 2016 Jul 30;18:176. doi: 10.1186/s13075-016-1073-3. PMID 27473164
- [Background] Perez de la Cruz S, Lambeck J. A new approach towards improved quality of life in fibromyalgia: a pilot study on the effects of an aquatic Ai Chi program. Int J Rheum Dis. 2018 Aug;21(8):1525-1532. doi: 10.1111/1756-185X.12930. Epub 2016 Jul 26. PMID 27457628
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Jones KD. Promoting physical activity in fibromyalgia. Pain Manag. 2016 May;6(4):321-4. doi: 10.2217/pmt-2016-0018. Epub 2016 Jun 17. No abstract available. PMID 27312858
- [Background] Okifuji A, Gao J, Bokat C, Hare BD. Management of fibromyalgia syndrome in 2016. Pain Manag. 2016 May;6(4):383-400. doi: 10.2217/pmt-2016-0006. Epub 2016 Jun 16. PMID 27306300
- [Background] Ericsson A, Mannerkorpi K. How to manage fatigue in fibromyalgia: nonpharmacological options. Pain Manag. 2016 May;6(4):331-8. doi: 10.2217/pmt-2016-0015. Epub 2016 Jun 14. PMID 27297077
- [Background] Ernberg M, Christidis N, Ghafouri B, Bileviciute-Ljungar I, Lofgren M, Larsson A, Palstam A, Bjersing J, Mannerkorpi K, Kosek E, Gerdle B. Effects of 15 weeks of resistance exercise on pro-inflammatory cytokine levels in the vastus lateralis muscle of patients with fibromyalgia. Arthritis Res Ther. 2016 Jun 13;18(1):137. doi: 10.1186/s13075-016-1041-y. PMID 27296860
- [Background] Bervoets DC, Luijsterburg PA, Alessie JJ, Buijs MJ, Verhagen AP. Massage therapy has short-term benefits for people with common musculoskeletal disorders compared to no treatment: a systematic review. J Physiother. 2015 Jul;61(3):106-16. doi: 10.1016/j.jphys.2015.05.018. Epub 2015 Jun 17. PMID 26093806
- [Background] Moustafa IM, Diab AA. The addition of upper cervical manipulative therapy in the treatment of patients with fibromyalgia: a randomized controlled trial. Rheumatol Int. 2015 Jul;35(7):1163-74. doi: 10.1007/s00296-015-3248-7. Epub 2015 Mar 18. PMID 25782585
- [Background] Yuan SL, Matsutani LA, Marques AP. Effectiveness of different styles of massage therapy in fibromyalgia: a systematic review and meta-analysis. Man Ther. 2015 Apr;20(2):257-64. doi: 10.1016/j.math.2014.09.003. Epub 2014 Oct 5. PMID 25457196
- [Background] Li YH, Wang FY, Feng CQ, Yang XF, Sun YH. Massage therapy for fibromyalgia: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2014 Feb 20;9(2):e89304. doi: 10.1371/journal.pone.0089304. eCollection 2014. PMID 24586677